CLINICAL TRIAL: NCT04573829
Title: PsyDoMa :Non-drug Approaches at Home for Alzheimer's Patients With Psycho-behavioural Disorders and Psycho-education for the Caregivers
Brief Title: PsyDoMa : Non-drug Approaches at Home for Alzheimer's Patients With Psycho-behavioural Disorders
Acronym: PSYDOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Fondation Mederic Alzheimer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-PP-19
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Behavioral Disorder
MeSH Terms: conditions — Mental Disorders | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-drug approaches at home (Experimental): Non-drug approaches at home three visits per week during six months and psycho-education for the caregivers one time per week for six months.
  Interventions: Procedure: Home visit

INTERVENTIONS:
Procedure: Home visit — Psychologist come once a week for the carer and three times a week for the patient

SUMMARY:
Recruitment is carried out directly at the geriatric unit of the CIMIEZ University Hospital Center by geriatric doctors during day consultation or in short stay unit. The doctor wil select carer -patient couples more likely to take part in the study. The investigator will give them an informative leaflet and they will have to sign the consent form.

A diagnosis is made by the investigator. The patient will first have to undergo a neurocognitive assessment carried out at the Cimiez Hospital (test for the evaluation of a cognitive deficit) by a psychologist.

The non-drug approaches presented will be carried out directly at the participant's home with the help of the carer for therapeutic purposes.

The therapeutic objectives and the choice of approaches are specified within the Personalised Accompaniment Project (PAP).

The carer, if he or she wishes, participates in the sessions in order to reproduce the behaviours implemented by the psychologist.

Different workshops will be offered : Cooking, Art Therapy, Games, Multi-sensory, Soft Gymnastic, Relaxation, Music and Reminisence.

Patients will received three visits per week during six months. The carer will receive one visit per week for six months.

ELIGIBILITY:
Inclusion Criteria:

For Patients

* Men or women over 65 years old showing signs of cognitive decline
* Living at home with specific needs ( meals, etc.) and the regular presence of a carer,
* Living in Nice
* Diagnosed with Alzheimer or dementia
* Presence of at least one behavioural disorder
* Person who agreed and signed the informed consent or his/her guardian For Carers
* Carer of the patient who meets the inclusion criteria: spouse, children, siblings or other family members at home or a professional carer.
* Person involved during the motivational interviewing session regarding the psychoeducational program.
* Person who agreed and signed the informed consent.

Exclusion Criteria:

For patients :

* Elderly person presenting no NINCDS- ADRDA criteria,
* Presence of sensory deficit (hearing or vision)
* Person unable to communicate,
* No regular presence of a home carer, waiting for a place in a nursing home
* Aging psychiatric pathologies,
* Elderly person attending a day-care centre

For carers :

* carer absent or not present enough,
* Elderly person with undiagnosed behavioural disorders
* Drug treatment that can interfere with assessments (psychotropic drugs, neuroleptics, etc.).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Ratio of personalised care projects completed | at the end of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, PU-PH, Principal Investigator — Nice University Hospital, Gerontology Department
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No